CLINICAL TRIAL: NCT00990119
Title: Vapotherm High Flow Therapy Via Nasal Cannula to Treat Respiratory Insufficiency in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: High Flow Therapy (HFT) to Treat Respiratory Insufficiency in Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot enrollment criteria did not yield intended population.
Sponsor: Vapotherm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRP-2009-03; Temple IRB protocol # 12573
Record Dates: First submitted 2009-08-27; First posted 2009-10-06 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency
Keywords: high flow therapy; high flow nasal cannula; chronic obstructive pulmonary disease; respiratory insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High FLow Therapy (Experimental): Use of High Flow Therapy for support of Respiratory Insufficiency
  Interventions: Device: Vapotherm High Flow Therapy
- NiPPV (Active Comparator)
  Interventions: Device: Non-invasive positive pressure ventilation

INTERVENTIONS:
Device: Vapotherm High Flow Therapy — use of high flow nasal cannula to support oxygenation and CO2 removal by flushing the nasopharynx with warmed, humidified respiratory gas at flow rates that exceed a patient's inspiratory flow rate
  Other Names: high flow nasal cannula
  Arms: High FLow Therapy
Device: Non-invasive positive pressure ventilation — Patients will be fit with an oronasal mask using a fitting gauge that will be applied by a respiratory therapist or other clinician skilled in management of NIPPV. Initial pressures will be at low end of suggested range but can be increased as rapidly as necessary to alleviate respiratory distress.
  Arms: NiPPV

SUMMARY:
The aim of this study is to see if the Vapotherm High Flow Therapy (HFT) device is effective to provide breathing support to patients with Chronic Obstructive Pulmonary Disease or COPD. The investigators believe that patients using HFT will not require as much use of therapies that provide pressure through a face mask, and are already recognized by FDA as support therapies for respiratory insufficiency.

DETAILED DESCRIPTION:
The overall objective of this study is to demonstrate that Vapotherm High Flow Therapy (HFT) via nasal cannula provides respiratory support to patients with COPD as a primary diagnosis, who present with respiratory insufficiency in the Emergency Department. We intend to demonstrate that Vapotherm HFT via nasal cannula will result in at least equivalent patient outcomes as the current standard of care, while eliminating the need for other non-invasive respiratory support devices cleared for the treatment of respiratory insufficiency. The current standard of care will include the use of other devices cleared by the FDA as respiratory assist devices for the treatment of adult respiratory insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Present to the Emergency Department with a history of COPD and with symptoms consistent with a diagnosis of respiratory insufficiency and exacerbation of COPD
* Must be hemodynamically stable as judged by treating clinician in the ED
* Primary complaint is shortness of breath, and presumed diagnosis is exacerbation of COPD

Exclusion Criteria:

* Fever
* Radiographic evidence of pneumonia
* Glasgow Coma score < 14 or unable to correctly answer at least one study-specific question

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Institution of positive pressure ventilation (PPV) or non-invasive positive pressure ventilation (NIPPV) | While in Emergency Department; at 24 hrs

SECONDARY OUTCOMES:
Borg Dyspnea Scale | 0, 2, 4 hrs
Respiratory Rate | 0, 2, 4 hrs
Arterial blood chemistry including pH, pCO2, pO2, HCO3-, BE- | 0, 2, 4 hrs
Pulse Ox and FIO2 | 0, 2, 4 hrs
Intensive Care Unit admission rate / Length of Stay | 7 days
Hospital Length of Stay | 7 days
Total duration of NIPPV/PPV or Vapotherm oxygen delivery | 7 days
Integrated FIO2 exposure | 7 days
Physician assessment - retractions, physician judgment of patient discomfort | 0, 2, 4 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Marla R Wolfson, PhD, Principal Investigator — Temple University; Nina Gentile, MD, Principal Investigator — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849